CLINICAL TRIAL: NCT00010426
Title: Randomized Study of New Formulation Ophthalmic Cysteamine Hydrochloride for Corneal Cystine Accumulation in Patients With Cystinosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Purpose: Treatment
Other Study IDs: 199/15704; SIGMATAU-FDR001769
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-04

CONDITIONS: Cystinosis
Keywords: cystinosis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Cystinosis; Rare Diseases; Urogenital Diseases | interventions — Cysteamine

INTERVENTIONS:
Drug: cysteamine hydrochloride

SUMMARY:
OBJECTIVES: I. Determine the proportion of patients with cystinosis who experience a serious adverse effect when treated with a new formulation of cysteamine hydrochloride for corneal cystine accumulation.

II. Determine the proportion of patients with a reduction in corneal crystal density of 1.00 unit when treated with this regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study Patients are randomized to receive the current formulation of cysteamine hydrochloride as drops in one eye and the new formulation of cysteamine hydrochloride as drops in the other eye.

Patients receive the two formulations of cysteamine hydrochloride in their assigned eyes every hour during waking hours daily for 6 months (safety study) or for 1 year (efficacy study).

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of cystinosis with more than 2 nmole half-cystine/mg protein in leukocytes OR presence of corneal crystals consistent with cystinosis and distributed in corneal stroma observed by slit lamp biomicroscopy
* Clinical history consistent with cystinosis
* Safety study: History of adherence with current eye drop and follow-up schedule on protocol #86-El-0062 Any crystal density score, including zero, on photographs, that has been stable or improved over the past year
* Efficacy study: Crystal density score at least 1.00 on photographs Concurrently on cysteamine for at least the past 6 months

--Prior/Concurrent Therapy--

* No prior cysteamine drops (efficacy study)

--Patient Characteristics--

* Age: 1 to 50 (safety study) 2 to 12 (efficacy study)
* Other: Willingness and ability to tolerate corneal photographs

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 1999-12; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. Lemanowicz, Study Chair — Leadiant Biosciences, Inc.